CLINICAL TRIAL: NCT04035434
Title: A Phase 1/2 Dose Escalation and Cohort Expansion Study of the Safety and Efficacy of Allogeneic CRISPR-Cas9-Engineered T Cells (CTX110) in Subjects With Relapsed or Refractory B-Cell Malignancies (CARBON)
Brief Title: A Safety and Efficacy Study Evaluating CTX110 in Subjects With Relapsed or Refractory B-Cell Malignancies (CARBON)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Patients to be followed up in the CRSP-ONC-LTF study
Sponsor: CRISPR Therapeutics AG (Industry)
Responsible Party: Sponsor
Organization: CRISPR Therapeutics (Industry)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CRSP-ONC-001
Record Dates: First submitted 2019-07-22; First posted 2019-07-29 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: B-cell Malignancy; Non-Hodgkin Lymphoma; B-cell Lymphoma; Adult B Cell ALL
Keywords: CAR T; Non-Hodgkin Lymphoma; NHL; Lymphoma; Allogeneic; Leukemia
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, B-Cell; Burkitt Lymphoma; Lymphoma; Leukemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- CTX110 (Experimental): Administered by IV infusion following lymphodepleting chemotherapy.
  Interventions: Biological: CTX110

INTERVENTIONS:
Biological: CTX110 — CTX110 (CD19-directed T-cell immunotherapy comprised of allogeneic T cells genetically modified ex vivo using CRISPR-Cas9 gene editing components

SUMMARY:
This is an open-label, multicenter, Phase 1/2 study evaluating the safety and efficacy of CTX110 in subjects with relapsed or refractory B-cell malignancies.

DETAILED DESCRIPTION:
The study may enroll up to 227 subjects in total. CTX110 is a CD19-directed chimeric antigen receptor (CAR) T cell immunotherapy comprised of allogeneic T cells prepared for the treatment of B cell malignancies. The cells are from healthy adult volunteer donors that are genetically modified ex vivo using CRISPR-Cas9 (clustered regularly interspaced short palindromic repeats/ CRISPR-associated protein 9) gene editing components (single guide RNA and Cas9 nuclease).

ELIGIBILITY:
Key Inclusion Criteria:

1. For NHL patients: Age ≥18 years. For B cell ALL patients: age ≥18 years to ≤70 years
2. Refractory or relapsed non-Hodgkin lymphoma, as evidenced by 2 or more lines of prior therapy, or histologically confirmed B cell ALL, refractory or relapsed.
3. Eastern Cooperative Oncology Group performance status 0 or 1.
4. Adequate renal, liver, cardiac and pulmonary organ function
5. Female subjects of childbearing potential and male subjects must agree to use acceptable method(s) of contraception from enrollment through at least 12 months after CTX110 infusion.

Key Exclusion Criteria:

1. For NHL patients: prior allogeneic HSCT. For B cell ALL patients: prior allogeneic HSCT within 6 months, and/or any evidence of GvHD.
2. History of central nervous system (CNS) involvement by malignancy
3. History of a seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
4. Presence of bacterial, viral, or fungal infection that is uncontrolled.
5. Positive for HIV, or active hepatitis B virus or hepatitis C virus infection.
6. Previous or concurrent malignancy, except basal cell or squamous cell skin carcinoma, adequately resected and in situ carcinoma of cervix, or a previous malignancy that was completely resected and has been in remission for ≥5 years.
7. For NHL patients: Use of systemic anti-tumor therapy or investigational agent within 14 days or 5 half-lives, whichever is longer, of CTX110 infusion. For B cell ALL patients: Use of systemic antitumor therapy within 7 days of CTX110 infusion.
8. Primary immunodeficiency disorder or active autoimmune disease requiring steroids and/or other immunosuppressive therapy.
9. Women who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2019-07-22 (Actual); Primary Completion 2024-10-04 (Actual); Study Completion 2024-10-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Annie Weaver, PhD, Study Director — CRISPR Therapeutics
Locations (33):
- United States (21):
  - Cedars Sinai, Los Angeles, California
  - UCSF Medical Center, San Francisco, California
  - Mayo Clinic, Jacksonville, Florida
  - Emory University Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago, Chicago, Illinois
  - University of Kansas, Westwood, Kansas
  - Markey Cancer Center, University of Kentucky, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Roswell Park Cancer Insitute, Buffalo, New York
  - Weill Cornell Medical College / New York Presbyterian Hospital, New York, New York
  - Duke University, Durham, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - Harold C. Simmons Comprehensive Cancer Center, UT Southwestern Medical Center, Dallas, Texas
  - Texas Transplant Institute, San Antonio, Texas
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - Peter MacCallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada
- France (3):
  - CHU de Lille, Lille
  - Institut Paoli-Calmettes, Marseille
  - Hôpital Saint Antoine, Paris
- Germany (2):
  - University of Hamburg, Hamburg
  - University Hospital Würzburg, Würzburg
- Spain (3):
  - Clinica Universidad de Navarra, Pamplona, Navarre
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario de Salamanca, Salamanca

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study comprises 4 cohorts: Cohorts A, B, and C enrolled adult participants with non-Hodgkin lymphoma (NHL); Cohort D enrolled participants with adult B cell acute lymphoblastic leukemia (ALL). A total of 93 participants were enrolled; 3 participants died prior to receiving CTX110 (1 due to pulmonary haemorrhage that occurred after lymphodepleting [LD] chemotherapy but was assessed as not related to LD chemotherapy, and 2 due to disease progression).
Pre-assignment Details: The study was designed to be divided into 2 phases. A total of 8 participants were enrolled in the Phase 2 dose expansion. Due to a high proportion of non-quantifiable values, the secondary efficacy endpoints for Phase 2 participants could not be calculated. The study was terminated early in Phase 2 at the sponsor's discretion.
Groups:
- Phase 1: NHL: Cohort A: Dose Level (DL) 1 (3×10^7 CAR+ T Cells): Participants with non-Hodgkin lymphoma (NHL) received lymphodepleting (LD) chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered intravenously (IV) once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 3x10^7 CAR+ T cells.
- Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 1x10^8 CAR+ T cells.
- Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 3×10^8 CAR+ T cells.
- Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 4.5×10^8 CAR+ T cells.
- Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells.
- Phase 1: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells); Phase 2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells and includes participants with 2 planned infusions during treatment course 1.
- Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (750 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells.
- Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells): Participants with NHL received daratumumab (16 mg/kg) at least 1 day before LD chemotherapy and within 10 days prior to CTX110 infusion. LD chemotherapy (fludarabine 30 mg/m² and cyclophosphamide 500 mg/m² IV daily for 3 days) was completed 48 hours to 7 days before CTX110 infusion. Participants with stable disease or better on Day 28 received additional daratumumab doses at Day 28 (±4 days) and Month 2 (±4 days). CTX110 was given as a single IV infusion of 3x10^8 CAR+ T cells.
- Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells): Participants with NHL received daratumumab (16 mg/kg) at least 1 day before LD chemotherapy and within 10 days prior to CTX110 infusion. LD chemotherapy (fludarabine 30 mg/m² and cyclophosphamide 500 mg/m² IV daily for 3 days) was completed 48 hours to 7 days before CTX110 infusion. Participants with stable disease or better on Day 28 received additional daratumumab doses at Day 28 (±4 days) and Month 2 (±4 days). CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells.
- Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells): Participants with B Cell ALL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 1x10^8 CAR+ T cells.
- Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells): Participants with B Cell ALL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 3×10^8 CAR+ T cells.
- Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells): Participants with B Cell ALL received daratumumab (16 mg/kg) at least 1 day before LD chemotherapy and within 10 days prior to CTX110 infusion. LD chemotherapy (fludarabine 30 mg/m² and cyclophosphamide 500 mg/m² IV daily for 3 days) was completed 48 hours to 7 days before CTX110 infusion. Participants with stable disease or better on Day 28 received additional daratumumab doses at Day 28 (±4 days) and Month 2 (±4 days). CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells.
Period: Dose Escalation Phase (Up to 5 Years)
Arm/Group | Phase 1: NHL: Cohort A: Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells)
Started | 3 | 3 | 6 | 6 | 10 | 4 | 0 | 1 | 5 | 5 | 4 | 5 | 7
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 6 | 6 | 10 | 4 | 0 | 1 | 5 | 5 | 4 | 5 | 7
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Death | 3 | 1 | 4 | 3 | 8 | 3 | 0 | 1 | 3 | 4 | 3 | 2 | 1
Not completed — Study terminated by the Sponsor | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 2 | 6
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Dose Expansion Phase (Up to 5 Years)
Arm/Group | Phase 1: NHL: Cohort A: Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells)
Started | 0 | 0 | 0 | 0 | 0 | 23 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 23 | 8 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 14 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Study terminated by the Sponsor | 0 | 0 | 0 | 0 | 0 | 8 | 4 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set: All participants who received CTX110 infusion.
Groups:
- Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells): Participants with non-Hodgkin lymphoma (NHL) received lymphodepleting (LD) chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered intravenously (IV) once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 3x10^7 CAR+ T cells.
- Cohort A: DL 2 (1x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 1x10^8 CAR+ T cells.
- Cohort A: DL 3 (3x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 3×10^8 CAR+ T cells.
- Cohort A: DL 3b (4.5x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 4.5×10^8 CAR+ T cells.
- Cohort A: DL 4a (6x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells.
- Cohort A: DL 4b (6x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells and includes participants with 2 planned infusions during treatment course 1.
- Cohort B: DL 4 (6x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (750 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells.
- Cohort C: DL 3 (3x10^8 CAR+ T Cells): Participants with NHL received daratumumab (16 mg/kg) at least 1 day before LD chemotherapy and within 10 days prior to CTX110 infusion. LD chemotherapy (fludarabine 30 mg/m² and cyclophosphamide 500 mg/m² IV daily for 3 days) was completed 48 hours to 7 days before CTX110 infusion. Participants with stable disease or better on Day 28 received additional daratumumab doses at Day 28 (±4 days) and Month 2 (±4 days). CTX110 was given as a single IV infusion of 3x10^8 CAR+ T cells.
- Cohort C: DL 4 (6x10^8 CAR+ T Cells): Participants with NHL received daratumumab (16 mg/kg) at least 1 day before LD chemotherapy and within 10 days prior to CTX110 infusion. LD chemotherapy (fludarabine 30 mg/m² and cyclophosphamide 500 mg/m² IV daily for 3 days) was completed 48 hours to 7 days before CTX110 infusion. Participants with stable disease or better on Day 28 received additional daratumumab doses at Day 28 (±4 days) and Month 2 (±4 days). CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells.
- B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells): Participants with B Cell ALL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 1x10^8 CAR+ T cells.
- B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells): Participants with B Cell ALL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 3×10^8 CAR+ T cells.
- B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells): Participants with B Cell ALL received daratumumab (16 mg/kg) at least 1 day before LD chemotherapy and within 10 days prior to CTX110 infusion. LD chemotherapy (fludarabine 30 mg/m² and cyclophosphamide 500 mg/m² IV daily for 3 days) was completed 48 hours to 7 days before CTX110 infusion. Participants with stable disease or better on Day 28 received additional daratumumab doses at Day 28 (±4 days) and Month 2 (±4 days). CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells.
- Total: Total of all reporting groups
Arm/Group | Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Cohort C: DL 4 (6x10^8 CAR+ T Cells) | B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) | B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) | B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells) | Total
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 10 | 35 | 1 | 5 | 5 | 4 | 5 | 7 | 90
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.3 (5.86) | 65.3 (8.08) | 68.2 (5.34) | 61.5 (18.29) | 61.8 (10.90) | 64.0 (11.74) | 59.0 (NA) — NA indicates standard deviation cannot be calculated for single participant | 71.0 (8.43) | 63.8 (6.65) | 35.0 (10.30) | 39.4 (13.83) | 47.7 (17.61) | 60.0 (14.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 4 | 2 | 2 | 9 | 0 | 2 | 2 | 1 | 2 | 3 | 29
  Male | 2 | 2 | 2 | 4 | 8 | 26 | 1 | 3 | 3 | 3 | 3 | 4 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 4
  White | 2 | 2 | 6 | 4 | 7 | 30 | 1 | 5 | 4 | 4 | 4 | 6 | 75
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 6

OUTCOME MEASURES:

1. Primary Outcome: Dose Escalation Phase 1: Number of Participants With Dose-limiting Toxicities (DLT) in NHL and B Cell ALL Population
Description: A DLT is defined as any of the following events occurring during the DLT evaluation period that persisted beyond the specified duration from onset: Grade ≥2 graft-versus-host disease (GvHD) that was steroid-refractory (e.g., progressive disease after 3 days of steroid treatment [e.g., 1 mg/kg/day], stable disease after 7 days, or partial response after 14 days of treatment); death during the DLT period, unless due to disease progression; Grade 4 neurotoxicity of any duration that was related or possibly related to CTX110; or any CTX110-related grade 3 or 4 toxicity deemed clinically significant by the investigator that did not improve within 72 hours.
Time Frame: Up to 28 days
Population: DLT Evaluable Set comprised of participants who received CTX110 and are followed for at least 28 days post-infusion or withdraw consent after experiencing a DLT.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells): Participants with non-Hodgkin lymphoma (NHL) received lymphodepleting (LD) chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered intravenously (IV) once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 3x10^7 CAR+ T cells.
- Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells): Participants with NHL received daratumumab (16 mg/kg) at least 1 day before LD chemotherapy and within 10 days prior to CTX110 infusion. LD chemotherapy (fludarabine 30 mg/m² and cyclophosphamide 500 mg/m² IV daily for 3 days) was completed 48 hours to 7 days before CTX110 infusion. Participants with stable disease or better on Day 28 received additional daratumumab doses at Day 28 (±4 days) and Month 2 (±4 days). CTX110 was given as a single IV infusion of 3*10^8 CAR+ T cells.
Arm/Group | Phase 1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 10 | 4 | 1 | 5 | 5 | 4 | 5 | 7
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Dose Expansion Phase 1 and Phase 2: Percentage of Participants With Objective Response Rate in NHL Population
Description: The objective response rate (complete response + partial response) was analyzed as per Lugano Response Criteria for Malignant Lymphoma, as determined by independent central radiology review. For participants who received the second course of treatment, the response assessments before and after the second course are combined for the derivation of objective response. Percentages are calculated with the number of participants in the specific analysis set in each column as the denominator. Confidence intervals (CI) of percentage are calculated with Clopper-Pearson exact method.
Time Frame: Up to 5 years
Population: Full Analysis Set comprised of participants who received CTX110 infusion have baseline and at least 1 post-baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Phase 1: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 23 | 8
Percentage of participants | 60.9 [38.5 to 80.3] | 75.0 [34.9 to 96.8]

3. Secondary Outcome: Dose Escalation Phase 1: Percentage of Participants With Objective Response Rate in B Cell ALL Population
Description: The objective response rate (complete response + complete remission with incomplete blood count recovery) was analyzed as per response criteria adapted from the National Comprehensive Cancer Network guidelines for treatment of acute lymphoblastic leukemia Version 2.2021, as determined by independent central radiology review. For -participants who receive the second course of treatment, the response assessments before and after the second course are combined for the derivation of objective response. Percentages are calculated with the number of participants in the specific analysis set in each column as the denominator. Confidence intervals (CI) of percentage are calculated with Clopper-Pearson exact method.
Time Frame: Up to 5 years
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 4 | 5 | 7
Percentage of Participants | 25.0 [0.6 to 80.6] | 40.0 [5.3 to 85.3] | 85.7 [42.1 to 99.6]

4. Secondary Outcome: Dose Escalation and Expansion Phase 1: Duration of Response in NHL Population
Description: Duration of response was only reported for the participants who showed objective response events. This was calculated as the time between first objective response and date of disease progression or death due to any cause. Median duration of response was calculated with the Kaplan-Meier method. Confidence intervals of median duration of response were calculated with the Brookmeyer and Crowley method with log-log transformation.
Time Frame: Up to 5 years
Population: Full Analysis Set: Participants who reported objective response events were analyzed. The duration of response for Phase 2 could not be calculated due to the high proportion of non-quantifiable values.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 0 | 1 | 4 | 4 | 7 | 16 | 1 | 3 | 2
Months |  | 9.20 [NA to NA] — Due to smaller number of events, 95% CI could not be calculated. | 3.75 [1.68 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 3.52 [0.95 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 1.02 [0.46 to 1.31] | 3.60 [1.91 to 8.57] | NA [NA to NA] — NA indicates single participant did not allow meaningful calculation of median and its 95% CI. | 2.20 [2.00 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 1.56 [1.05 to NA] — Due to smaller number of events, upper 95% CI could not be calculated.

5. Secondary Outcome: Dose Escalation and Expansion Phase 1: Progression Free Survival (PFS) in NHL Population
Description: Progression-free survival (PFS) and event-free survival were calculated as the difference between date of CTX110 infusion and date of disease progression or death due to any cause. The median of PFS was calculated with the Kaplan-Meier method. The CIs of median PFS were calculated with the Brookmeyer and Crowley method with log-log transformation.
Time Frame: Up to 5 years
Population: Full Analysis Set: Participants who reported PFS events were analyzed. The progression free survival for Phase 2 could not be calculated due to the high proportion of non-quantifiable values.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 10 | 27 | 1 | 5 | 5
Months | 0.92 [0.79 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 1.91 [0.85 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 2.43 [0.95 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 1.54 [0.82 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 1.77 [0.76 to 2.10] | 2.83 [1.02 to 3.94] | NA [NA to NA] — NA indicates single participant did not allow meaningful calculation of median and its 95% CI. | 2.92 [0.79 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 1.94 [0.92 to NA] — Due to smaller number of events, upper 95% CI could not be calculated.

6. Secondary Outcome: Dose Escalation and Expansion Phase 1: Median Overall Survival (OS) in NHL Population
Description: Overall survival was calculated as the time between date of first dose of CTX110 and death due to any cause. Participants who are alive at the data cutoff date will be censored at their last date known to be alive. Median overall survival was calculated with the Kaplan-Meier method. CIs of median overall survival were calculated with the Brookmeyer and Crowley method with log-log transformation.
Time Frame: Up to 5 years
Population: Full Analysis Set: Participants reporting overall survival rate were analyzed. The median overall survival for Phase 2 could not be calculated due to the high proportion of non-quantifiable values.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Phase 1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 10 | 27 | 1 | 5 | 5
Months | 5.03 [2.73 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 37.16 [1.05 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 7.77 [2.96 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | NA [1.61 to NA] — Due to smaller number of events, the median and upper 95% CI could not be calculated. | 5.16 [1.71 to 27.73] | 14.26 [4.47 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 12.12 [NA to NA] — Due to smaller number of events, 95% CI could not be calculated. | 7.39 [1.18 to NA] — Due to smaller number of events, upper 95% CI could not be calculated. | 7.62 [1.71 to NA] — Due to smaller number of events, upper 95% CI could not be calculated.

7. Secondary Outcome: Dose Escalation and Expansion: Number of Participants With Treatment Emergent Adverse Events (TEAEs) in NHL and B Cell ALL Population
Description: A TEAE was any untoward medical occurrence or worsening of a pre-existing condition in a clinical trial participant who received the investigational medicinal product, regardless of a causal relationship with the treatment. An AE had to be classified as a serious adverse event (SAE) if it resulted in death, was life-threatening, required or prolonged hospitalization, caused persistent or significant disability or incapacity, led to a congenital anomaly or birth defect in a newborn, or was deemed a significant medical event by the investigator based on medical judgment.
Time Frame: Up to 5 years
Population: Safety Analysis Set. The safety data are presented by treatment received and not by study phase.
Measure: Count of Participants; unit: Participants
Groups:
- Phase1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells): Participants with non-Hodgkin lymphoma (NHL) received lymphodepleting (LD) chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered intravenously (IV) once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 3x10^7 CAR+ T cells.
- Phase 1/2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells and includes participants with 2 planned infusions during treatment course 1.
- Phase 1: Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells): Participants with NHL received daratumumab (16 mg/kg) at least 1 day before LD chemotherapy and within 10 days prior to CTX110 infusion. LD chemotherapy (fludarabine 30 mg/m² and cyclophosphamide 500 mg/m² IV daily for 3 days) was completed 48 hours to 7 days before CTX110 infusion. Participants with stable disease or better on Day 28 received additional daratumumab doses at Day 28 (±4 days) and Month 2 (±4 days). CTX110 was given as a single IV infusion of 3x10^8 CAR+ T cells.
Arm/Group | Phase1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Phase 1/2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 10 | 35 | 1 | 5 | 5 | 4 | 5 | 7
Participants | 3 | 3 | 6 | 6 | 10 | 34 | 1 | 5 | 5 | 4 | 5 | 7

8. Secondary Outcome: Dose Escalation and Expansion: Number of Participants With Clinically Significant Laboratory Abnormalities in NHL and B Cell ALL Population
Description: Blood samples were collected for the analysis of laboratory parameters including hematology, clinical chemistry and coagulation parameters. The hematology parameters included: Lymphocyte count decreased, Neutrophil count decreased, White blood cell decreased, Anemia, Platelet count decreased, leukocytosis and Lymphocyte count increased. Chemistry parameters included: Hypoalbuminemia, Aspartate aminotransferase increased, Alanine aminotransferase increased, Hypokalemia, Chronic kidney disease, Blood bilirubin increased, Creatinine increased, Hypermagnesemia, Hypernatremia, Hypercalcemia, Hyperkalemia, and Hypoglycemia. Coagulation parameters included: Activated partial thromboplastin time prolonged, Fibrinogen decreased, and INR increased. Grade 3 and above severity of laboratory abnormalities are considered as clinically significant laboratory abnormalities.
Time Frame: Up to 5 years
Population: Safety Analysis Set. The safety data are presented by treatment received and not by study phase.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells): B Cell ALL: Cohort D: DL 3 (3*10^8 CAR+ T Cells) Participants with B Cell ALL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 3×10^8 CAR+ T cells.
Arm/Group | Phase 1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Phase 1/2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 10 | 35 | 1 | 5 | 5 | 4 | 5 | 7
Participants
  Lymphocyte count decreased | 3 | 3 | 6 | 6 | 10 | 35 | 1 | 5 | 5 | 4 | 5 | 7
  Neutrophil count decreased | 3 | 3 | 6 | 6 | 10 | 35 | 1 | 5 | 5 | 4 | 5 | 7
  White blood cell decreased | 3 | 2 | 6 | 6 | 10 | 35 | 1 | 5 | 5 | 4 | 5 | 7
  Anemia | 1 | 1 | 4 | 3 | 8 | 17 | 0 | 2 | 3 | 2 | 3 | 3
  Platelet count decreased | 1 | 2 | 3 | 4 | 6 | 19 | 1 | 2 | 5 | 2 | 3 | 3
  Lymphocyte count increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Hypoalbuminemia | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
  Aspartate aminotransferase increased | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1
  Alanine aminotransferase increased | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 0 | 2
  Hypokalemia | 1 | 1 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
  Hypercalcemia | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0
  Hyperkalemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
  Chronic kidney disease | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Blood bilirubin increased | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Creatinine increased | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Hypernatremia | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Activated partial thromboplastin time prolonged | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 1 | 1 | 1 | 1 | 0
  Fibrinogen decreased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  INR increased | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Leukocytosis | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

9. Secondary Outcome: Dose Escalation and Expansion: Mean Concentration of CTX110 in Blood Over Time Following the First CTX110 Infusion in NHL Population
Description: Blood samples were collected for the analysis of mean concentration of CTX110 in blood (copies per micrograms deoxyribose nucleic acid [DNA]) over time following the first CTX110 infusion. Cohort A DL4a and DL4b were combined, as the same dose was administered. Mean concentration values of CTX110 have been presented by dose level.
Time Frame: Day 1 pre-infusion, Day 1 post-infusion, Day 2, Day 3, Day 5, Day 8, Day 10, Day 14, Day 21, Day 28, Month 2, Month 3, Month 6, Month 9, Month 12 and Month 24
Population: Full Analysis Set. Only those participants with data available at specified timepoints has been presented.
Measure: Mean (Standard Deviation); unit: Copies per micrograms DNA
Groups:
- Phase 1/2: NHL: Cohort A: DL 4a + DL 4b(6x10^8 CAR+ T Cells): Participants with NHL received LD chemotherapy consisting of fludarabine (30 mg/m²) and cyclophosphamide (500 mg/m²) administered IV once daily for three consecutive days. LD chemotherapy was completed at least 48 hours, but no more than 7 days, before infusion of CTX110. CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells. Cohort A DL4a and DL4b were combined for pharmacokinetic analysis as same dose of CTX110 was administered
Arm/Group | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells) | Phase 1/2: NHL: Cohort A: DL 4a + DL 4b(6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 6 | 6 | 1 | 5 | 5 | 45
Copies per micrograms DNA
  Day 1 pre-infusion: number analyzed (Participants) | 3 | 6 | 1 | 2 | 3 | 43
  Day 1 pre-infusion | 2.90 (0.000) | 3.55 (1.592) | 2.90 (NA) — The standard deviation cannot be calculated for single participant | 2.90 (0.000) | 2.90 (0.000) | 3.08 (0.934)
  Day 1 post-infusion: number analyzed (Participants) | 2 | 6 | 1 | 2 | 4 | 42
  Day 1 post-infusion | 144.95 (147.856) | 829.37 (1552.483) | 472.20 (NA) — The standard deviation cannot be calculated for single participant | 105.22 (23.028) | 636.29 (352.700) | 979.25 (1658.499)
  Day 2: number analyzed (Participants) | 4 | 6 | 1 | 3 | 4 | 42
  Day 2 | 7.27 (6.403) | 10.77 (13.999) | 28.57 (NA) — The standard deviation cannot be calculated for single participant | 35.62 (22.359) | 72.39 (107.323) | 42.39 (101.461)
  Day 3: number analyzed (Participants) | 4 | 6 | 1 | 3 | 3 | 39
  Day 3 | 8.36 (5.310) | 12.46 (9.656) | 22.03 (NA) — The standard deviation cannot be calculated for single participant | 16.76 (13.050) | 204.43 (300.219) | 35.80 (98.739)
  Day 5: number analyzed (Participants) | 4 | 3 | 1 | 4 | 4 | 38
  Day 5 | 25.47 (21.898) | 220.78 (246.411) | 311.67 (NA) — The standard deviation cannot be calculated for single participant | 80.40 (33.878) | 487.13 (262.303) | 770.14 (3312.713)
  Day 8: number analyzed (Participants) | 5 | 6 | 1 | 3 | 2 | 39
  Day 8 | 3763.68 (8138.642) | 4337.42 (7721.088) | 13269.43 (NA) — The standard deviation cannot be calculated for single participant | 5844.98 (9600.631) | 719.13 (231.318) | 10277.87 (27526.126)
  Day 10: number analyzed (Participants) | 4 | 5 | 1 | 5 | 5 | 39
  Day 10 | 180.87 (209.131) | 452.03 (941.853) | 25719.13 (NA) — The standard deviation cannot be calculated for single participant | 19018.53 (42303.294) | 297.91 (248.623) | 4056.03 (19737.607)
  Day 14: number analyzed (Participants) | 4 | 6 | 1 | 5 | 4 | 40
  Day 14 | 2.90 (0.000) | 3.55 (1.592) | 9.93 (NA) — The standard deviation cannot be calculated for single participant | 2435.23 (5423.525) | 51.73 (87.882) | 2186.81 (13766.282)
  Day 21: number analyzed (Participants) | 4 | 6 | 1 | 4 | 4 | 41
  Day 21 | 2.90 (0.000) | 2.90 (0.000) | 2.90 (NA) — The standard deviation cannot be calculated for single participant | 64.48 (123.167) | 3.88 (1.950) | 2537.64 (11074.754)
  Day 28: number analyzed (Participants) | 5 | 5 | 1 | 5 | 4 | 37
  Day 28 | 4.00 (2.452) | 2.90 (0.000) | 2.90 (NA) — The standard deviation cannot be calculated for single participant | 6.67 (8.437) | 2.90 (NA) — The standard deviation cannot be calculated for single participant | 8.32 (28.058)
  Month 2: number analyzed (Participants) | 2 | 2 | 1 | 3 | 1 | 5
  Month 2 | 3.88 (1.379) | 2.90 (0.000) | NA (NA) — Mean and standard deviation could not be calculated as all concentration values were below the lower limit of quantification | 11.17 (14.318) | 2.90 (NA) — The standard deviation cannot be calculated for single participant | 2.90 (0.000)
  Month 3: number analyzed (Participants) | 3 | 2 | 1 | 3 | 1 | 1
  Month 3 | 3.55 (1.126) | 2.90 (0.000) | NA (NA) — Mean and standard deviation could not be calculated as all concentration values were below the lower limit of quantification | 2.90 (0.000) | 2.90 (NA) — The standard deviation cannot be calculated for single participant | 2.90 (NA) — The standard deviation cannot be calculated for single participant
  Month 6: number analyzed (Participants) | 2 | 1 | 1 | 0 | 0 | 0
  Month 6 | 2.90 (0.000) | 2.90 (NA) — The standard deviation cannot be calculated for single participant | NA (NA) — Mean and standard deviation could not be calculated as all concentration values were below the lower limit of quantification |  |  |
  Month 9: number analyzed (Participants) | 0 | 1 | 1 | 0 | 0 | 0
  Month 9 |  | 2.90 (NA) — The standard deviation cannot be calculated for single participant | NA (NA) — Mean and standard deviation could not be calculated as all concentration values were below the lower limit of quantification |  |  |
  Month 12: number analyzed (Participants) | 0 | 1 | 1 | 5 | 1 | 0
  Month 12 |  | 2.90 (NA) — The standard deviation cannot be calculated for single participant | NA (NA) — Mean and standard deviation could not be calculated as all concentration values were below the lower limit of quantification | 2.90 (NA) — The standard deviation cannot be calculated for single participant | 2.90 (NA) — The standard deviation cannot be calculated for single participant |
  Month 24: number analyzed (Participants) | 0 | 1 | 1 | 5 | 5 | 0
  Month 24 |  | 2.90 (NA) — The standard deviation cannot be calculated for single participant | NA (NA) — Mean and standard deviation could not be calculated as all concentration values were below the lower limit of quantification | NA (NA) — Mean and standard deviation could not be calculated as all concentration values were below the lower limit of quantification | NA (NA) — Mean and standard deviation could not be calculated as all concentration values were below the lower limit of quantification |

10. Secondary Outcome: Dose Escalation and Expansion Phase 1: Mean Concentration of CTX110 in Blood Over Time Following the First CTX110 Infusion in B Cell ALL Population
Description: Blood samples were collected for the analysis of mean concentration of CTX110 in blood (copies per micrograms deoxyribose nucleic acid [DNA]) over time following the first CTX110 infusion.
Time Frame: Day 1 pre-infusion, Day 1 post-infusion, Day 2, Day 3, Day 5, Day 8, Day 10, Day 14, Day 21, Day 28, and Month 2
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: Copies per micrograms DNA
Groups:
- Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells): B Cell ALL: Cohort D: DL 4 (6*10^8 CAR+ T Cells) Participants with B Cell ALL received daratumumab (16 mg/kg) at least 1 day before LD chemotherapy and within 10 days prior to CTX110 infusion. LD chemotherapy (fludarabine 30 mg/m² and cyclophosphamide 500 mg/m² IV daily for 3 days) was completed 48 hours to 7 days before CTX110 infusion. Participants with stable disease or better on Day 28 received additional daratumumab doses at Day 28 (±4 days) and Month 2 (±4 days). CTX110 was given as a single IV infusion of 6×10^8 CAR+ T cells.
Arm/Group | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 4 | 5 | 7
Copies per micrograms DNA
  Day 1 pre-infusion: number analyzed (Participants) | 4 | 5 | 4
  Day 1 pre-infusion | 13.43 (21.067) | 3.29 (0.872) | 2.90 (0.000)
  Day 1 post-infusion: number analyzed (Participants) | 4 | 5 | 4
  Day 1 post-infusion | 781.86 (1395.907) | 1983.57 (1677.746) | 602.75 (521.357)
  Day 2: number analyzed (Participants) | 3 | 4 | 6
  Day 2 | 4.20 (2.252) | 93.47 (149.220) | 18.13 (17.532)
  Day 3: number analyzed (Participants) | 3 | 4 | 6
  Day 3 | 13.46 (14.905) | 20.47 (25.356) | 7.95 (4.705)
  Day 5: number analyzed (Participants) | 3 | 4 | 6
  Day 5 | 28.65 (36.011) | 42.37 (47.444) | 62.85 (124.743)
  Day 8: number analyzed (Participants) | 4 | 4 | 6
  Day 8 | 71.30 (118.215) | 16846.17 (33459.507) | 15941.89 (30200.959)
  Day 10: number analyzed (Participants) | 3 | 4 | 6
  Day 10 | 226.32 (290.508) | 26.17 (41.517) | 14177.59 (23256.089)
  Day 14: number analyzed (Participants) | 2 | 4 | 6
  Day 14 | 1040.13 (1466.869) | 2.90 (0.000) | 380.29 (924.424)
  Day 21: number analyzed (Participants) | 3 | 4 | 7
  Day 21 | 3.55 (1.126) | 2.90 (0.000) | 2.90 (0.000)
  Day 28: number analyzed (Participants) | 2 | 4 | 6
  Day 28 | 2.90 (0.000) | 2.90 (0.000) | 2.90 (0.000)
  Month 2: number analyzed (Participants) | 1 | 1 | 1
  Month 2 | 2.90 (NA) — The standard deviation cannot be calculated for single participant | 2.90 (NA) — The standard deviation cannot be calculated for single participant | 2.90 (NA) — The standard deviation cannot be calculated for single participant

11. Secondary Outcome: Dose Escalation and Expansion: Number of Participants With Serious Adverse Events (SAEs) in NHL and B Cell ALL Population
Description: An AE had to be classified as a serious adverse event (SAE) if it resulted in death, was life-threatening, required or prolonged hospitalization, caused persistent or significant disability or incapacity, led to a congenital anomaly or birth defect in a newborn, or was deemed a significant medical event by the investigator based on medical judgment.
Time Frame: Up to 5 years
Population: Safety Analysis Set. The safety data are presented by treatment received and not by study phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Phase 1/2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells)
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 10 | 35 | 1 | 5 | 5 | 4 | 5 | 7
Participants | 3 | 2 | 1 | 1 | 5 | 8 | 0 | 1 | 4 | 3 | 3 | 1

ADVERSE EVENTS:
Time Frame: Up to 5 years
Description: The safety analysis set is comprised of all participants who are enrolled and received study treatment. The participants in the safety analysis set were classified according to the received study treatment. The safety analysis set was the default set for safety analyses.
Arm/Group | Phase 1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) | Phase 1/2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells)
All-Cause Mortality (participants affected / at risk) | 3/3 | 2/3 | 4/11 | 3/6 | 9/10 | 21/35 | 1/1 | 3/5 | 4/5 | 4/4 | 2/5 | 1/7
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/3 | 1/6 | 1/6 | 5/10 | 8/35 | 0/1 | 1/5 | 4/5 | 3/4 | 3/5 | 1/7
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 6/6 | 10/10 | 34/35 | 1/1 | 5/5 | 5/5 | 4/4 | 5/5 | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) (N=3) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) (N=3) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) (N=6) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) (N=6) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) (N=10) | Phase 1/2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) (N=35) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) (N=1) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) (N=5) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells) (N=5) | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) (N=4) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) (N=5) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells) (N=7)
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 2 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertensive encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 1 | 1 | 1 | 3 | 3 | 0 | 0 | 2 | 0 | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Enterococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Escherichia sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pseudomonal sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Venoocclusive liver disease (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Facial paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: NHL: Cohort A Dose Level (DL) 1 (3×10^7 CAR+ T Cells) (N=3) | Phase 1: NHL: Cohort A: DL 2 (1x10^8 CAR+ T Cells) (N=3) | Phase 1: NHL: Cohort A: DL 3 (3x10^8 CAR+ T Cells) (N=6) | Phase 1: NHL: Cohort A: DL 3b (4.5x10^8 CAR+ T Cells) (N=6) | Phase 1: NHL: Cohort A: DL 4a (6x10^8 CAR+ T Cells) (N=10) | Phase 1/2: NHL: Cohort A: DL 4b (6x10^8 CAR+ T Cells) (N=35) | Phase 1: NHL: Cohort B: DL 4 (6x10^8 CAR+ T Cells) (N=1) | Phase 1: NHL: Cohort C: DL 3 (3x10^8 CAR+ T Cells) (N=5) | Phase 1: NHL: Cohort C: DL 4 (6x10^8 CAR+ T Cells) (N=5) | Phase 1: B Cell ALL: Cohort D: DL 2 (1x10^8 CAR+ T Cells) (N=4) | Phase 1: B Cell ALL: Cohort D: DL 3 (3x10^8 CAR+ T Cells) (N=5) | Phase 1: B Cell ALL: Cohort D: DL 4 (6x10^8 CAR+ T Cells) (N=7)
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1 | 0 | 3 | 9 | 0 | 0 | 0 | 1 | 0 | 4
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1 | 0 | 5 | 0 | 1 | 0 | 0 | 1 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0
Catheter site pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Feeling abnormal (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 1 | 1 | 1 | 2 | 4 | 16 | 1 | 2 | 1 | 0 | 3 | 5
Hypogammaglobulinaemia (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Genital cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 4 | 1 | 0 | 1 | 0 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1 | 2 | 2 | 0 | 2 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Hallucination, auditory (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac murmur (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 1 | 1 | 3 | 4 | 0 | 0 | 1 | 1 | 1 | 2
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Anosmia (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysarthria (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasticity (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 2 | 5 | 3 | 8 | 20 | 0 | 2 | 4 | 1 | 3 | 6
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 3 | 3 | 7 | 16 | 0 | 1 | 3 | 0 | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 2 | 5 | 3 | 5 | 12 | 0 | 1 | 3 | 0 | 2 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 2 | 0 | 2 | 11 | 1 | 3 | 4 | 2 | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0
Methaemoglobinaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lymph node pain (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitreous haemorrhage (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 3 | 1 | 1 | 10 | 0 | 1 | 0 | 1 | 1 | 3
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 2 | 9 | 1 | 2 | 1 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 2 | 0 | 7 | 0 | 2 | 2 | 1 | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 2 | 0 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 2 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hepatic vascular thrombosis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 2 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory syncytial virus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia moraxella (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Viruria (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bacterial disease carrier (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinovirus infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 2 | 2 | 3 | 1 | 1 | 1 | 1 | 1 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 0 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperchloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypervolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Magnesium deficiency (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site swelling (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 3
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Catheter site thrombosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Graft versus host disease (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Clostridium difficile infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 1 | 2 | 3 | 0 | 0 | 1 | 1 | 0 | 0
CD4 lymphocytes decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Lymph node palpable (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Respiratory syncytial virus test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis haemorrhagic (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Limitations of the trial such as small numbers of participants analysed or technical problems leading to unreliable data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/34/NCT04035434/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-16): https://cdn.clinicaltrials.gov/large-docs/34/NCT04035434/SAP_001.pdf